CLINICAL TRIAL: NCT06579001
Title: Effect of Nasal Spray Dexmedetomidine on Emergence Delirium Prevention in Total Hip Replacement in the Elderly Under General Anesthesia: a Randomized Clinical Trial
Brief Title: Effect of Nasal Spray Dexmedetomidine on Emergence Delirium Prevention in Total Hip Replacement
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2024-0592
Record Dates: First submitted 2024-08-11; First posted 2024-08-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-07

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dex group (Experimental): at least 20 min before the introduction of anesthesia, the patient takes the sitting position, the head is slightly tilted forward, and the product is kept upright. Insert the nostril at the same Angle as the nasal cavity. Press down on the spray pump evenly with the index and middle fingers at the same time, and press the pump to the bottom at one time for 1 spray (25ug). After 1 spray on both nostrils, tilt your head back slightly and inhale gently. After staying for about 30 s, 1 spray was applied to each nostril on both sides for a total of 4 sprays (100ug).
  Interventions: Drug: Nasal spray dexmedetomidine
- Saline group (Placebo Comparator): Normal saline packaged in the same appearance was used
  Interventions: Drug: Nasal spray dexmedetomidine

INTERVENTIONS:
Drug: Nasal spray dexmedetomidine — Nasal spray dexmedetomidine or saline was used 100ug per patient acording to the group assignment
  Other Names: saline

SUMMARY:
Emergence Delirium (ED) is a common postoperative complication refers to an acute brain dysfunction that occurs during the recovery from general anesthesia, which is mainly characterized by sudden attention and consciousness disorders. The occurrence of ED increases the risk of self-injury, wound dehiscence, accidental catheter dislocation, and postoperative delirium, and is also associated with postoperative cognitive deterioration and increased utilization of medical resources after discharge.

DETAILED DESCRIPTION:
The incidence of hip fracture after surgery in patients over 55 years old is about 45%, and ED is highly predictive of delirium during postoperative hospitalization, which occurs in about 1/3 of ED patients during postoperative hospitalization.

It has been suggested that if delirium is monitored only on the first postoperative day and not at the PACU stage, up to 53% of delirium cases may be missed.

Studies have shown that perioperative application of dexmedetomidine can reduce the risk of postoperative delirium to a certain extent. However, intravenous dexmedetomidine usually leads to problems with delayed extubation, residual sedation, and prolonged PACU stay.

Previous studies have shown that intranasal dexmedetomidine improves perioperative sleep quality and neurocognitive deficits in elderly patients undergoing laparoscopic gynecologic surgery. Compared with intravenous administration, intranasal administration of dexmedetomidine resulted in milder hemodynamic fluctuations. However, stable nasal spray bioavailability is superior to intravenous dosage forms for nasal use.

Based on the above background, this study aims to investigate the effect of nasal spray of dexmedetomidine on the prevention of emergence delirium after total hip replacement in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years old
2. Total hip arthroplasty under general anesthesia
3. ASA II-III
4. Informed consent was obtained from patients or their guardians

Exclusion Criteria:

1. Allergy or contraindication to dexmedetomidine
2. Severe rhinitis and nasal deformity
3. Severe bradycardia (heart rate <50 beats/minute) or atrioventricular block of grade 2 or higher, permanent pacemaker implantation, severe heart failure or ejection fraction <30%
4. Patients with previous myocardial infarction, unstable angina pectoris, severe arrhythmia, and cardiac insufficiency
5. Emergency surgery
6. Severe hepatic and renal dysfunction (Child-Pugh class B and C, CKD3-5)
7. Preoperative mental illness, cognitive impairment, and communication difficulties could not be evaluated in the study
8. Preoperative delirium was present

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-08 (Estimated)

PRIMARY OUTCOMES:
emergency delirium | postoperative
  RASS&CAM-ICU, delirium was judged according to whether there were positive features in the questionnaire

SECONDARY OUTCOMES:
Preoperative anxiety score | preoperative
  Perioperative anxiety scale，PAS-7, score range: 0-28, higher score means more anxiety
Postoperative delirium | postoperative 3 days
  3D-CAM,delirium was judged according to whether there were positive features in the questionnaire
time to extubation | postoperative 3 days
  time to extubation
PACU stay | postoperative 3 days
  length of PACU stay
Hemodynamic changes | introperative
  between drug administration and anesthesia introduction
PONV | postoperative 3 days
  the incidence of nausea and /or vomiting
sleep quality | postoperative 3 days
  RCSQ, 0-100, higher score means higher sleep quality
Pain score | postoperative 3 days
  NRS, 0-10, 0 means no pain, 10 means severe pain

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 闗闗, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No